CLINICAL TRIAL: NCT05034614
Title: Pap Smear Collection With the Papette Brush: A Pragmatic Study
Brief Title: Pap Smear Collection With the Papette Brush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Danielle J. O'Laughlin, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-006131
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Cervical Cancer Screening
Keywords: Pap Smear Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pap smears using the Papette (Other): Papette brush used to collect a Pap smear sample as standard of care.
  Interventions: Diagnostic Test: Papette brush collection
- Pap smears using the traditional spatula/cytology brush (Other): Spatula/cytology brush used to collect a Pap smear sample as standard of care.
  Interventions: Diagnostic Test: Spatula/cytology brush collection

INTERVENTIONS:
Diagnostic Test: Papette brush collection — Cervical cell brush that gathers collects cervical cells during Pap smear collection
  Arms: Pap smears using the Papette
Diagnostic Test: Spatula/cytology brush collection — Combination of extended-tip spatula with endocervical brush that collects cervical cells during Pap smear collection
  Arms: Pap smears using the traditional spatula/cytology brush

SUMMARY:
This research study is comparing Pap smear collection techniques using the Papette brush to traditional spatula and cytology brush for cervical cancer screening

DETAILED DESCRIPTION:
At the investigators institution the investigators have been using both the traditional spatula and cytology and the Papette brush for Pap smear collection. The investigators will be comparing adequacy of sample rates, provider perceived pain and bleeding and overall satisfaction with each collection technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult women, aged 21-64 years old.
* Have given consent for medical records to be accessed.
* Who will have a Pap smear exam in CIM from July 2021 through June 2022.

Exclusion Criteria:

* Women, age < 21 or > 64.
* Has vaginal spotting present during cervical sampling.
* Did not give consent to have medical records accessed.

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 756 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle O'Laughlin, PA-C, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pap Smears Using the Papette | Pap Smears Using the Traditional Spatula/Cytology Brush
Started | 357 | 399
Completed | 357 | 399
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pap Smears Using the Papette | Pap Smears Using the Traditional Spatula/Cytology Brush | Total
Number analyzed (Participants) | 357 | 399 | 756
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (13.64) | 46.8 (12.34) | 45.4 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 357 | 399 | 756
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 0 | 1 | 1
  Asian | 17 | 28 | 45
  Black or African American | 13 | 16 | 29
  Other | 17 | 16 | 33
  White | 309 | 334 | 643
  Unknown | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 357 | 399 | 756

OUTCOME MEASURES:

1. Primary Outcome: Specimen Adequacy
Description: Number of subjects who's samples have cervical cellular adequacy for a satisfactory evaluation indicated on the cytology report
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Pap Smears Using the Papette | Pap Smears Using the Traditional Spatula/Cytology Brush
Number analyzed (Participants) | 357 | 399
Participants | 335 | 371
Statistical Analysis 1: Comparison: Pap Smears Using the Papette vs Pap Smears Using the Traditional Spatula/Cytology Brush; Test type: Superiority; p = .75, Chi-squared

2. Secondary Outcome: Cervical Bleeding With Collection
Description: Number of subjects to experience bleeding with collection of samples during the Pap smear exam
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Pap Smears Using the Papette | Pap Smears Using the Traditional Spatula/Cytology Brush
Number analyzed (Participants) | 357 | 399
Participants | 0 | 0

3. Secondary Outcome: Collection Time
Description: The amount of time it takes to collect a sample measured in seconds
Time Frame: Baseline
Population: Data was not collected or analyzed for this outcome measure
Arm/Group | Pap Smears Using the Papette | Pap Smears Using the Traditional Spatula/Cytology Brush
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Perceived Pain
Description: Provider-reported survey to assess patient perceived pain for Papette brush compare to spatula/cytology bush technic as more, the same, or less patient perceived pain.
Time Frame: Baseline
Population: Data was not collected nor analyzed
Arm/Group | Pap Smears Using the Papette | Pap Smears Using the Traditional Spatula/Cytology Brush
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all subjects from baseline to end of study for approximately 1 hour
Arm/Group | Pap Smears Using the Papette | Pap Smears Using the Traditional Spatula/Cytology Brush
All-Cause Mortality (participants affected / at risk) | 0/357 | 0/399
Serious Adverse Events (participants affected / at risk) | 0/357 | 0/399
Other Adverse Events (participants affected / at risk) | 0/357 | 0/399

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT05034614/Prot_SAP_000.pdf